CLINICAL TRIAL: NCT07300709
Title: Renal Histopathology and Transcriptomic Analysis in Hepatorenal Syndrome During Liver Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Tiffany Cho-Lam Wong, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UW25-392
Record Dates: First submitted 2025-10-02; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hepatorenal Syndrome, Liver Regeneration; AKI - Acute Kidney Injury; Liver Transplant
Keywords: Hepatorenal syndrome; HRS; HRS AKI; acute kidney injury; liver transplant; renal biopsy; renal histopathology; transcriptomics
MeSH Terms: conditions — Hepatorenal Syndrome; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal biopsy (Experimental): To examine the actual structural changes in kidneys of patients with HRS through tissue biopsy and advanced molecular analysis, and hope that may help us better understand the disease mechanism and potentially improve treatment approaches
  Interventions: Procedure: renal biopsy

INTERVENTIONS:
Procedure: renal biopsy — To examine the actual structural changes in kidneys of patients with HRS through tissue biopsy and advanced molecular analysis, and hope that may help us better understand the disease mechanism and potentially improve treatment approaches

SUMMARY:
Hepatorenal Syndrome (HRS) is a serious complication that can occur in patients with liver cirrhosis, characterised by kidney dysfunction, or acute kidney failure (AKI). While it has traditionally been thought that HRS affects structurally normal kidneys and is completely reversible with liver transplantation, recent evidence suggests this may not always be the case.

The purpose of this study is to examine the actual structural changes in the kidneys of patients with HRS through tissue biopsy and advanced molecular analysis. This may help us better understand the disease mechanism and potentially improve treatment approaches. We aim to challenge the current understanding that HRS always occurs in structurally normal kidneys and is always reversible after liver transplantation. This study will provide valuable insights into the pathophysiology of HRS and may lead to improved diagnostic and treatment strategies in the future.

This is a 3-year single center prospective, non-randomised, open label study at Queen Mary Hospital, The University of Hong Kong. All consecutive patients accepted on the liver transplant waiting list will be invited to participate. Patient will undergo several procedures related to liver transplant and kidney assessment, and receive liver transplantation and renal biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be able to understand and provide informed consent
2. Age ≥ 18 years of age at time of study entry
3. Accepted for liver transplantation (LT)
4. Fulfill the diagnostic criteria of HRS AKI according to International Club of Ascites (ICA) guidelines

3-month post transplant renal biopsy inclusion criteria:

1. Patient with adequate intraoperative renal biopsy
2. Patient must be able to understand and provide informed consent

Exclusion Criteria:

1. Inability or unwillingness to give written informed consent
2. Patient with known pre-existing renal disease
3. Patient with solitary kidney
4. Re-transplantation
5. ABO-incompatible LT
6. Fail to provide 3-month post transplant renal biopsy

3-month post transplant renal biopsy exclusion criteria:

1. Graft failure after LT
2. Any condition deemed inappropriate by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with HRS AKI | up to 3 years
  Proportion of patients with HRS AKI who have normal, reversible or permanent injury on renal histopathology
Histopathological changes | up to 3 years
  Histopathological changes and their association with clinical parameters

SECONDARY OUTCOMES:
Duration of HRS AKI | up to 3 years
  Incidence and duration of HRS AKI
Response to standard treatment (Terlipressin and albumin) | up to 3 years
  Response to standard treatment (Terlipressin and albumin)
Perioperative morbidity | up to 3 years
  Perioperative morbidity including need and duration for renal replacement therapy
Post-transplant renal recovery rates | up to 3 years
  Post-transplant renal recovery rates
Transcriptomic signature differences | up to 3 years
  Transcriptomic signature differences between HRS AKI and non-HRS AKI patients

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT07300709/Prot_SAP_000.pdf